CLINICAL TRIAL: NCT00436085
Title: Randomized Controlled Trial of Stress Management Training in Individuals With HIV Infection
Brief Title: Randomized Controlled Trial of Stress Management Training in HIV
Acronym: SWISSIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3346C0-100907
Record Dates: First submitted 2007-02-15; First posted 2007-02-16 (Estimated); Last update posted 2007-02-16 (Estimated); Status verified 2007-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Behavioral: Cognitive behavioral stress management training

SUMMARY:
The introduction of highly active antiretroviral therapy (HAART) has dramatically changed the consequences of an HIV infection, which is now viewed as a chronic disease. As in other chronic diseases, emotional distress and depressive symptoms are highly prevalent in HIV-infected patients. Psychological factors such as these have been associated with lower quality of life, lower adherence to therapy and also with a higher risk for mortality and disease progression. Psychosocial interventions, such as group-based cognitive behavioral stress management (CBSM) training, have been shown to reduce distress and psychological symptoms in HIV-infected patients. These psychosocial effects are paralleled by changes in physiological parameters, such as cortisol, DHEA-S, testosterones, catecholamines, and naïve T-cell counts. While these results are congruent with recent evidence of the interaction between psychological, neuroendocrine and immunological parameters in HIV-infected patients, it needs to be shown whether the reported effects hold true in the HAART era. Most importantly, it also needs to be ascertained whether these interventions have an impact on immunological and virological HIV parameters as well as on mortality and morbidity in HIV patients. We propose a randomized controlled one-year prospective evaluation of a group-based CBSM training in 80 HIV-infected patients. Participating patients will be recruited at cooperating centers of the Swiss HIV Cohort Study and randomly assigned to CBSM training or waiting control group condition. At baseline, post-training and two follow-up (6 and 12 months) assessments, effects of the CBSM on psychological, physiological and clinical out-come variables in HIV-infected patients under HAART will be evaluated. Additionally, the effects of CBSM on the neuroendocrine and autonomic stress reactivity in HIV-infected patients will be assessed, thus evaluating a possible direct pathway between emotional distress and physiological HIV-relevant parameters. In conclusion, the planned research project evaluates the effectiveness of a standardized psychosocial intervention as a possible component of a comprehensive disease management in HIV-infected patients under HAART.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 65 years of age
* Sufficient German-speaking abilities to participate in group therapy
* cARTwithin the previous three months,
* CD4 lymphocyte count above 100 cells/mL

Exclusion Criteria:

* Active opportunistic infection at baseline
* Formal psychotherapy within the previous three months
* Intravenous drug users
* Diagnosable current major psychiatric disorder (bipolar affective disorder, psychotic disorders, major depression with melancholia) and diagnosis of antisocial and borderline personality disorders at baseline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-12; Study Completion 2005-12

PRIMARY OUTCOMES:
CD4 cell count
HIV viral load

SECONDARY OUTCOMES:
Depression and Anxiety
QUality of life

CONTACTS AND LOCATIONS:
Overall Officials: Jens Gaab, PhD, Principal Investigator — Clinical Psychology and PSychotherapy, Institute of Psychology, University of Zürich; Rainer Weber, MD, Principal Investigator — University Hospital, Zürich; Ulrike Ehlert, PhD, Principal Investigator — Clinical Psychology and Psychotherapy, Institute of Psychology, University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland